CLINICAL TRIAL: NCT02287805
Title: Craniosynostosis: How to Improve the Diagnosis and Assist Patients and Their Families?
Brief Title: Qualitative and Quantitative Study Which Aims to Determine the Specifics of the Announcement for the Diagnosis of Patients With Craniosynostosis and Their Parents to Better Support Them in Their Care
Acronym: AmAc
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Université de Cergy Pontoise (Unknown)
Responsible Party: Sponsor
Other Study IDs: URC 1073
Record Dates: First submitted 2014-10-10; First posted 2014-11-11 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Craniosynostosis
Keywords: craniosynostosis; simple form; complex form; diagnostic; announcement; impacts
MeSH Terms: conditions — Craniosynostoses; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- quantitative survey 1: parents of 300 patients with craniosynostosis diagnostic
  Interventions: Other: quantitative survey
- qualitative survey: * parents of 12 newly diagnosed patients, they will be seen 3 times (after the diagnosis, 3 months after surgery, 1 year after surgery
  * 12 patients aged over 15 years, operated more than 10 years before
  Interventions: Other: qualitative survey
- quantitative survey 2: * 100 parents of patients 1 year after surgery
  * 100 parents of patients, 5 years after the operation
  * 100 patients aged over 15 years and operated over 10 years ago
  Interventions: Other: quantitative survey

INTERVENTIONS:
Other: qualitative survey
  Groups: qualitative survey
Other: quantitative survey
  Groups: quantitative survey 1; quantitative survey 2

SUMMARY:
The purposes of this study are:

* to better understand the experience of the announcement for the diagnostic of craniosynostosis to patients and their families to improve the understanding of it and it modes of appropriation
* to compare the announcement process concerning "simple" and "complex" forms.
* to identify the intra-family issues at the announcement of a genetic mutation.
* to reconstruct the care course of patients by analyzing the time of the announcement and the post-operative period.

DETAILED DESCRIPTION:
The supported hypothesis is that the diagnosis of craniosynostosis disturbs the initial family pattern. The different forms of the disease will have different repercussions on intra-family relationships.

The quality of the announcement done by the doctor influences the way how the subjects (parents and patients themselves) appropriate and incorporate it at short, medium and long term.

This research will contribute to the knowledge of this rare disease by different scientific communities: social sciences, medicine and neuropsychology. The originality of this research lies in interdisciplinary teams involved and the cross looks between professional and associative fields.

To better understand the impact of congenital malformations and specifically those related to craniosynostosis, the experiences of children and their families at short, medium and long term, the research will take place in the center of reference "Dysostoses craniofacial", Pediatric Neurosurgery Service at the Necker Hospital in Paris.

Prior to fieldwork, a thorough literature search will be conducted on issues related to our subject: the announcement, psychological, identity, family and social impacts, as well as the specifics of the disease and its manifestations.

The fieldwork will be included in a longitudinal approach which will be located at the intersection of quantitative and qualitative methods.

ELIGIBILITY:
Inclusion Criteria :

Group 1 :

Parents of operated children with a clinical diagnosis of craniosynostosis

Group 2 :

* Parents of newly diagnosed children for a craniosynostosis who will be operated
* Children aged 15 who were operated for a craniosynostosis at least 10 years ago

Group 3 :

* Parents of newly diagnosed children for a craniosynostosis who will be operated
* Children aged 15 who were operated for a craniosynostosis at least 10 years ago

Exclusion Criteria:

* nothing to declare

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children with craniosynostosis who are followed by the Reference Center "Dysostoses craniofaciales" and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 574 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
measure by questionnaire the conditions and experiences of the announcement concerning craniosynostosis (simple or complex) | 5 months
  Analysis of the questionnaires will permit us to learn more about the conditions and experiences of the announcement concerning different profiles families whose experience has been received differently depending on the type of craniosynostosis (simple or complex), the medical history or sociodemographic characteristics.

SECONDARY OUTCOMES:
measure by interview the conditions and experiences of the announcement concerning craniosynostosis (simple or complex) interview | 16 months
  In a longitudinal perspective, we will develop interview guides. For conducting interviews, we will use the life story method. The interest of the life story is that it provides a method to study the modes of appropriation of the announcement and the way in which subjects incorporate it into their life history.
measure by an other questionnaire the conditions and experiences of the announcement concerning craniosynostosis (simple or complex) | 6 months
  From the results of all the interviews (from qualitative survey) and the analysis of questionnaires from the quantitative survey 1, we will develop questionnaires for themes and issues that have emerged from those analyses (accompanying the announcement of genetic mutation in the family, aesthetics, education ...). It will then develop targeted questionnaires, based on the analysis of interviews and questionnaires from the quantitative survey. The goal will be a deepening of themes.

CONTACTS AND LOCATIONS:
Overall Officials: Séverine Colinet, PhD, Study Chair — Cergy University
Locations (1):
- Centre de référence des dysostoses craniofaciales, Hôpital Necker Enfants Malades, Paris, France